CLINICAL TRIAL: NCT00002725
Title: PHASE II EVALUATION OF BRYOSTATIN-1 (NSC 339555) IN NON-HODGKIN'S LYMPHOMA
Brief Title: Bryostatin-1 in Treating Patients With Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02239; MDA-DM-95061; NCI-T95-0035D; CDR0000064591 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-23 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2000-10

CONDITIONS: Lymphoma
Keywords: recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — bryostatin 1; Drug Therapy

ARMS (1):
- Arm I (Experimental): Single-Agent Chemotherapy/Differentiation Therapy. Bryostatin 1, BRYO, NSC-339555.
  Interventions: Drug: bryostatin 1; Drug: chemotherapy

INTERVENTIONS:
Drug: bryostatin 1
Drug: chemotherapy

SUMMARY:
Phase II trial to study the effectiveness of bryostatin-1 in treating patients with recurrent non-Hodgkin's lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response to bryostatin 1 (BRYO) administered weekly for 3 weeks in patients with relapsed non-Hodgkin's lymphoma.

II. Assess the toxic effects of this treatment. III. Establish the correlation between PKC isoenzyme activity and BRYO function in lymphoma cells and normal lymphocytes.

IV. Determine the pharmacokinetic profile of BRYO and its relationship to pharmacodynamics.

OUTLINE:

Single-Agent Chemotherapy/Differentiation Therapy. Bryostatin 1, BRYO, NSC-339555.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma
* Working formulation low-, intermediate-, and high-grade histologies eligible
* Mantle cell and marginal zone lymphoma eligible
* Relapse after at least 1 doxorubicin-containing regimen required
* No more than 2 prior chemotherapy regimens
* One prior biologic therapy in addition to the 2 prior chemotherapy regimens allowed
* No prior bone marrow transplantation
* Ineligible for treatment on higher priority protocols
* Patients eligible for bone marrow transplantation may be treated to reduce tumor bulk
* Bidimensionally measurable disease required
* No history of primary or metastatic CNS disease

PATIENT CHARACTERISTICS:

* Age: Any age
* Performance status: Zubrod 0-2
* Life expectancy: Greater than 12 weeks
* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.8 mg/dL
* Transaminases no greater than 2.5 times normal
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance greater than 70 mL/min
* No HIV antibody
* No serious intercurrent illness
* No pregnant or nursing women
* Effective contraception required of fertile patients throughout study and for 1 year thereafter

PRIOR CONCURRENT THERAPY:

-At least 4 weeks since prior therapy (6 weeks since mitomycin) and recovered

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1996-08; Primary Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Romaguera, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States